CLINICAL TRIAL: NCT03464604
Title: Melanoma Accuracy Study, Phase Two
Brief Title: Melanoma Accuracy Study; Phase 2
Status: Terminated | Type: Observational
Why Stopped: COVID forced the termination of this study. No impact on participants already enrolled.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 1023029
Record Dates: First submitted 2018-02-27; First posted 2018-03-14 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 Control group: Patients randomized into this group will follow normal standard of care in Nova Scotia
- Group 2 Active group: Patients randomized into this group will be part of the active arm of the study. They will be pre-screened and asked the following questions:
  1. Sign an Information and Authorization form
  2. Demographic data: gender, date of birth, ethnicity
  3. Health history (duration of lesion, changes in lesion, specific changes, who identified the lesion, measurement in two greatest dimensions radially and color.
  Interventions: Diagnostic Test: active

INTERVENTIONS:
Diagnostic Test: active — Pre-screening for melanoma by qualified nurse
  Groups: Group 2 Active group

SUMMARY:
The purpose of this study is to evaluate the process, accuracy and patient outcomes of pre-screening dermatology referrals in a clinical setting by a qualified nurse. The long-range goal of the proposed program is to improve referral wait times for patients to see a dermatologist for lesions suspicious for melanoma in comparison to normal standards of care in NS. If effective, this screening program would decrease wait times for those patients with lesions suspicious for melanoma providing earlier diagnosis and expedited treatment, and potentially reducing mortality rates.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the process, accuracy and patient outcomes of pre-screening dermatology referrals in a clinical setting by a qualified nurse using a dermatoscope, triaging suspicious lesions vs. benign lesions. The long-range goal of the proposed program is to improve referral wait times for patients to see a dermatologist for lesions suspicious for melanoma in comparison to normal standards of care in NS. If effective, this screening program would decrease wait times for those patients with lesions suspicious for melanoma providing earlier diagnosis and expedited treatment, and potentially reducing mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* New referral from a general practitioner to a dermatologist
* Males and females, over the age of 18 are eligible to participate
* Written informed consent from the patient
* Lesion or mole is new, changing color, growing rapidly or has a change in sensation
* Willing to have the lesion excised if necessary per standard of care
* Ability to complete the imaging procedure and willing to complete a basic history
* Pigmented lesion considered low, moderate or high risk for melanoma by a general practitioner

Exclusion Criteria

* Lesions which are not amenable
* Participant unable to read, understand or sign consent
* Participant under active care by a dermatologist
* Lesion <2 mm or >15mm in diameter
* Lesion located on areas of scars, crusts, psoriasis, eczema or similar skin conditions
* Lesion on hair covered areas (e.g. scalp, beard, mustache) where hair cannot be removed
* Lesions located on genitalia not accessible to equipment
* Lesions located in an area that has previously biopsied or subjected to any kind of surgical or ablative procedure
* Lesion with foreign matter, e.g. tattoo or splinter
* Lesion and/or reference located on acute sunburn
* Skin surface not measurable, e.g. lesion on a stalk
* Skin surface not accessible, e.g. inside ears, ears, under nails
* Skin not intact (measurement area), e.g. bleeding or with clinically noticeable ulceration
* Lesions located within 1cm of the eye
* Lesions light in pigment or thick and nodular
* Participants not willing to have the lesion excised

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are 18+ (male or female) referred to the Department of Dermatology at the NSHA for a suspicious pigmented lesion(s).
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Pre-screening lesions low to moderate risk for melanoma by a nurse, will facilitate a more timely diagnosis of melanoma. | 3 years
  Pre-screening referrals to the Department of Dermatology by a qualified nurse for patients with lesions, low to moderate risk for melanoma, would facilitate a more timely diagnosis of melanoma, and appropriate triaging of benign lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Lngley, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No